CLINICAL TRIAL: NCT01034592
Title: A Pilot Study of Lenalidomide in Adult Diamond-Blackfan Anemia Patients With Red Blood Cell Transfusion-Dependent Anemia
Brief Title: Pilot Lenalidomide in Adult Diamond-Blackfan Anemia Patients w/ RBC Transfusion-Dependent Anemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual related to rarity of Diamond-Blackfan anemia (DBA)
Sponsor: Jason Robert Gotlib (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jason Robert Gotlib, Prof-Med Ctr Line in Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-16822; SU-12082009-4523 (Other: Stanford University); RV-0365 (Other: Celgene Corporation); HEMMDS0022 (Other: OnCore)
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Anemia; Leukemia; Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Anemia; Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Subjects will initially receive lenalidomide 2.5 mg, and may escalate up to 2.5 mg/wk up to 5 mg 3x/wk, depending toxicity and response.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 2.5 mg/wk up to 5 mg 3x/wk
  Other Names: Revlimid; CC-5013

SUMMARY:
This is a single-center, single arm, open-label study of oral lenalidomide monotherapy administered to red blood cell (RBC) transfusion dependent adult subjects with Diamond-Blackfan Anemia (DBA).

Primary Objective: To evaluate the erythroid response rate as measured by rate of red blood cell transfusion independence [MDS International Working Group (IWG) 2000 Criteria will be applied].

Secondary Objective: 1)To evaluate the tolerability and safety profile of lenalidomide in patients with DBA and other inherited marrow failure syndromes 2) To correlate response to lenalidomide with biologic surrogates of DBA including ribosomal protein mutation status, ex vivo erythroid colony growth, and microarray gene expression

DETAILED DESCRIPTION:
This pilot study will utilize an intra-patient dose escalation design. Cycles are 28 days in length. Subjects will receive lenalidomide 2.5 mg weekly during days 1 to 21 of cycle 1 (dose level 1). If patients do not experience any grade > 3 hematologic or non-hematologic toxicity, the dose will be increased to 2.5 mg twice weekly on days 1 to 21 of cycle 2 (dose level 2). If patients do not experience any grade > 3 hematologic or non-hematologic toxicity, the dose will be increased to 5 mg twice weekly on days 1 to 21 of cycle 3 (dose level 3). If patients do not experience any grade >3 hematologic or non-hematologic toxicity, the dose will be increased to 5 mg thrice weekly on days 1 to 21 of cycle 4 (dose level 4). Patients who experience grade >3 hematologic or non-hematologic toxicity at dose level 1 will be discontinued from study. Patients who experience grade > 3 hematologic or non-hematologic toxicity at dose level 2, 3, or 4 will have the lenalidomide held and dose reduced according to protocol dose interruption/modification algorithms (section 5.5.3). If at least a minor erythroid response is not achieved at the end of 8 cycles of treatment, patients will be discontinued from study. If a minor or major erythroid response is achieved after completion of 8 cycles of treatment, patients can continue study drug on a maintenance phase until loss of erythroid response (return to baseline hemoglobin or transfusion requirement) or unacceptable toxicity.

ELIGIBILITY:
INCLUSION CRITERIA

* Understand and voluntarily sign an informed consent form
* Diagnosis of DBA
* Age ≥ 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Red blood cell transfusion-dependent with a requirement of at least one unit of RBCs per month for the 2 months prior to study enrollment (eg, 2 units/8 weeks)
* If applicable, ongoing therapy with a stable or decreasing dose of prednisone ≤ 60 mg/d or corticosteroid equivalent, for which there has been no treatment-related improvement in RBC transfusion requirements for at least 2 months prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry.
* Laboratory test results within these ranges:

  * Absolute neutrophil count (ANC) ≥ 1500/uL
  * Platelet (Plt) count ≥ 100,000/uL
  * Serum creatinine ≤ 2.0 mg/dL
  * Direct bilirubin ≤ 1.5 mg/dL
  * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Disease-free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of ≥ 50 milli-International Units (MIU)/mL within 10 to 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Able to take aspirin (81 to 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin)

EXCLUSION CRITERIA

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy (excluding steroids) specifically used for DBA within 28 days of baseline including metoclopramide, leucine, danazol, or other hormonal therapy
* Clinically significant anemia due to factors such as iron, B12, folate deficiencies, autoimmune or hereditary hemolysis, or gastrointestinal bleeding.
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or infectious hepatitis, type A, B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robert Gotlib, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell (RBC) Transfusion Independence
Description: Red blood cell (RBC) transfusion independence is reported as the number of subjects who achieve a continuous absence of the intravenous infusion of any RBC transfusion during any consecutive "rolling" 56 days during the treatment period.
Time Frame: 6 months
Population: All treated subjects were analyzed.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
participants | 0

2. Secondary Outcome: Red Blood Cell (RBC) Transfusions
Description: The effect on red blood cell (RBC) transfusions was assessed as the number of participants that achieved a greater than 50% decrease in RBC transfusion requirements.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Hemoglobin Concentration
Description: The effect on hemoglobin concentration was assessed as the change from baseline, measured in g/dL.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
g/dL | 0.4 [0.4 to 0.4]

4. Secondary Outcome: Neutrophil Response
Description: The effect on neutrophil levels was assessed as the change in neutrophil count from baseline.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis.
Measure: Median (Full Range); unit: 1000/uL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
1000/uL | 0.50 [0.10 to 0.91]

5. Secondary Outcome: Platelet Response
Description: The effect on platelet levels as assessed as the change in platelet count from baseline.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis.
Measure: Median (Full Range); unit: 1000/uL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
1000/uL | 25.5 [-20.0 to 71.0]

6. Secondary Outcome: Duration of Response
Description: The response duration was measured from the last of the consecutive 56 days during which the subject was free of red blood cells (RBC) transfusions to the date of the first RBC transfusion after the 56-day RBC-transfusion-free period.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis, but never demonstrated any therapeutic response.
Measure: Median (Full Range); unit: days
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
days | 0 [0 to 0]

7. Secondary Outcome: Toxicity
Description: Toxicity was assessed as the number of adverse events related to lenalidomide.
Time Frame: 6 months
Population: Both participants were assessed and contributed to the analysis.
Measure: Number; unit: Related Adverse Events
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
Related Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the treatment and maintenance phase of the study, for a total of 2 years.
Groups:
- Serious Adverse Events: Serious Adverse Events include: adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, result in a persistent or significant disability/incapacity or result in a congenital anomaly/birth defect. Other important medical events, based upon appropriate medical judgment, may also be considered Serious Adverse Events if a trial participant's health is at risk and intervention is required to prevent an outcome mentioned.
Arm/Group | Serious Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serious Adverse Events (N=2)
Fatigue (General disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase, increased (Investigations) | 1 (1)
Alanine aminotransferase, increased (Investigations) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 2 subjects were enrolled on this protocol. Low accrual was related to various factors. Given the accrual status, no substantive conclusions about the efficacy or safety of lenalidomide in adults with Diamond-Blackfan Anemia could be reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No